CLINICAL TRIAL: NCT04451954
Title: Safety and Immunogenicity of Quadrivalent Recombinant Influenza Vaccine Formulations Containing Different H3 Hemagglutinin Antigens Without or With Adjuvant in Healthy Adult Subjects
Brief Title: Study of Recombinant Influenza Vaccine Containing Different H3 Antigens Without or With Adjuvant in Healthy Adult Subjects
Acronym: FBP00004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FBP00004; U1111-1239-0391 (Other: UTN)
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunisation; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1: Quadrivalent RIV with H3 strain 1, without adjuvant (Experimental): 1 injection of quadrivalent RIV containing H3 strain 1, without adjuvant, in participants ≥ 50 years old
  Interventions: Biological: Quadrivalent RIV with H3 strain 1
- Group 2: Quadrivalent RIV with H3 strain 1, with adjuvant (Experimental): 1 injection of quadrivalent RIV containing H3 strain 1, with adjuvant, in participants ≥ 50 years old
  Interventions: Biological: Quadrivalent RIV with H3 strain 1 and adjuvant
- Group 3: Quadrivalent RIV with H3 strain 2, without adjuvant (Experimental): 1 injection of quadrivalent RIV containing H3 strain 2, without adjuvant, in participants ≥ 50 years old
  Interventions: Biological: Quadrivalent RIV with H3 strain 2
- Group 4: Quadrivalent RIV with H3 strain 2, with adjuvant (Experimental): 1 injection of quadrivalent RIV containing H3 strain 2, with adjuvant, in participants ≥ 50 years old
  Interventions: Biological: Quadrivalent RIV with H3 strain 2 and adjuvant
- Group 5: Quadrivalent RIV Control, without adjuvant (Active Comparator): 1 injection of quadrivalent RIV containing 2018-19 Northern Hemisphere (NH) recommended H3 strain, without adjuvant, in participants ≥ 50 years old
  Interventions: Biological: Quadrivalent RIV with 2018-2019 NH H3 strain
- Group 6: Quadrivalent RIV Control, with adjuvant (Active Comparator): 1 injection of quadrivalent RIV containing 2018-19 NH recommended H3 strain, with adjuvant, in participants ≥ 50 years old
  Interventions: Biological: Quadrivalent RIV with 2018-2019 NH H3 strain and adjuvant
- Group 7: Quadrivalent RIV Control, without adjuvant (Active Comparator): 1 injection of quadrivalent RIV containing 2018-19 NH recommended H3 strain, without adjuvant, in participants 18-30 years old
  Interventions: Biological: Quadrivalent RIV with 2018-2019 NH H3 strain

INTERVENTIONS:
Biological: Quadrivalent RIV with H3 strain 1 — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Group 1: Quadrivalent RIV with H3 strain 1, without adjuvant
Biological: Quadrivalent RIV with H3 strain 1 and adjuvant — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Group 2: Quadrivalent RIV with H3 strain 1, with adjuvant
Biological: Quadrivalent RIV with H3 strain 2 — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Group 3: Quadrivalent RIV with H3 strain 2, without adjuvant
Biological: Quadrivalent RIV with H3 strain 2 and adjuvant — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Group 4: Quadrivalent RIV with H3 strain 2, with adjuvant
Biological: Quadrivalent RIV with 2018-2019 NH H3 strain — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Group 5: Quadrivalent RIV Control, without adjuvant; Group 7: Quadrivalent RIV Control, without adjuvant
Biological: Quadrivalent RIV with 2018-2019 NH H3 strain and adjuvant — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Group 6: Quadrivalent RIV Control, with adjuvant

SUMMARY:
The primary objectives of the study are:

* To describe the safety profile of the different formulations in all participants
* To describe the hemagglutinin inhibition (HAI) and seroneutralization (SN) antibody responses against hemagglutinin (H1, H3, B/Victoria, and B/Yamagata) antigens present in the control vaccine in all groups at all timepoints.

The secondary objectives are:

* To describe antigenic coverage in each group by assessing the HAI and SN antibody responses against a panel of H3 antigens (not present in any of the vaccine formulations).
* To describe SN antibody responses in each group against each of the H3 antigens.
* To compare H3 HAI and SN antibody responses for the groups with quadrivalent recombinant influenza vaccine (RIV) formulations with H3 antigens to those of the quadrivalent RIV control group.
* To compare the HAI and SN antibody responses for the groups with quadrivalent RIV formulation with adjuvant to the group without adjuvant.

DETAILED DESCRIPTION:
Study duration per participant is approximately 1 year

ELIGIBILITY:
Inclusion criteria :

* Older adults: Aged 50 years and older on the day of inclusion Young adults: Aged 18 to 30 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion criteria:

* Participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 12 weeks postvaccination. To be considered of non-childbearing potential, a female must be premenarche, or postmenopausal for at least 1 year, or surgically sterile
* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following study vaccination
* Previous vaccination against influenza during either of the previous 2 influenza seasons (2018-2019 and 2019-2020) with any licensed or investigational influenza vaccine
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; immunosuppressive therapy (such as anticancer chemotherapy or radiation therapy, within the preceding 6 months); or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months) or receipt of hydroxychloroquine within the preceding 4 weeks
* Dementia or any other cognitive condition at a stage that could interfere with following the trial procedures
* Have known active or recently active (12 months) neoplastic disease or a history of any hematologic malignancy
* History of influenza infection during either of the previous 2 influenza seasons (2018- 2019 or 2019-2020), confirmed by laboratory tests (including rapid tests) at that time
* History of laboratory confirmed coronavirus disease 2019 (COVID-19), confirmed with a nucleic acid amplification test on a respiratory specimen, or known exposure to severe acute respiratory syndrome coronavirus (SARS-CoV-2) positive confirmed close contact (eg, family member, housemate, daycare provider, aged parent requiring care), in the 30 days preceding vaccination, at the discretion of the investigator
* Self-reported or documented seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances
* Have any diagnosis, current or past, of an autoimmune disease
* Thrombocytopenia or bleeding disorder, contraindicating intramuscular vaccination based on investigator's judgment
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Any change in chronic prescription medication or change in medication dose or dosage in the 60 days prior to enrollment
* Alcohol abuse or substance abuse that, in the opinion of the investigator, might interfere with the study conduct or completion
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Any current or past diagnosis of chronic pulmonary disease including asthma (history of childhood asthma is allowed), cystic fibrosis and chronic pulmonary obstructive disease
* Have taken a high-dose inhaled corticosteroid within 6 months prior to study vaccination
* Body mass index of 40 or higher
* Any current or past diagnosis of cardiac disease (eg, coronary artery disease, heart failure, or valvular heart disease [mild mitral valve prolapse allowed]). Participants with isolated primary (essential) hypertension are allowed
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (oral temperature ≥100.4 F [≥38.0 C]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an investigator or employee of the investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the investigator or employee with direct involvement in the proposed study
* Personal or family history of Guillain-Barré syndrome
* History of chronic kidney disease
* Current or past diagnosis of thyroid disease (eg, thyroiditis [including Hashimoto's thyroiditis], hyperthyroidism, and hypothyroidism)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events | Within 30 minutes after vaccination
  Immediate adverse events are unsolicited systemic adverse events reported in the 30 minutes after vaccination
Number of participants with solicited injection site or systemic reactions | From Day 0 to Day 7
  Solicited injection site reactions: injection site pain, erythema, swelling, induration and bruising; solicited systemic reactions: fever, headache, malaise, and myalgia
Number of participants with unsolicited adverse events | From Day 0 to Day 28
  Unsolicited (spontaneously reported) adverse events not not fulfilling criteria for solicited reactions
Number of participants with serious adverse events | From Day 0 to Day 365
  Serious adverse events are collected throughout the study
Number of participants with adverse events of special interest | From Day 0 to Day 365
  Adverse events of special interest are collected throughout the study
Clinical safety laboratory test results | From Day 0 to Day 7
  Laboratory tests include complete blood count (CBC), platelet count, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, serum creatinine, serum lipase, and serum amylase)
HAI and SN antibody titers against influenza antigens in the quadrivalent RIV control vaccine | From Day 0 to Day 365
  Influenza antibody titers are measured by HAI and SN assays
Individual HAI and SN titers ratio against influenza antigens in the quadrivalent RIV control vaccine | From Day 0 to Day 90
  Titers ratio is calculated for the following time points: Day 7/Day 0, Day 28/Day 0, and Day 90/Day 0
Number of participants with seroconversion to influenza antigens in the quadrivalent RIV control vaccine | From Day 0 to Day 28
  Seroconversion is defined as HAI antibody titer < 10 [1/dil] at Day 0 and post-injection titer ≥ 40 [1/dil] at Day 28, or titer ≥ 10 [1/dil] at Day 0 and a ≥ 4-fold increase in titer [1/dil] at Day 28)
HAI Ab titer ≥ 40 [1/dil] | From Day 0 to Day 365
  Influenza vaccine antibody titers are measured by HAI assay
2-fold and 4-fold increase in SN titers | From Day 0 to Day 28
  Influenza vaccine antibody titers are measured by SN assay

SECONDARY OUTCOMES:
HAI antibody titers against influenza H3 antigens not present in the vaccine formulations and the SN antibody titers against each of the H3 antigens | Day 0, Day 7, Day 28, Day 90, Day 180, and Day 365
  Influenza vaccine antibody titers are measured by HAI and SN assays
Individual HAI titer ratios against influenza H3 antigens not present in the vaccine formulations and individual SN titer ratio against each of the H3 antigens | From Day 0 to Day 90
  Titer ratio is calculated for the following time points: Day 7/Day 0, Day 28/Day 0, Day 90/Day 0
Number of participants with seroconversion to influenza H3 antigens not present in the vaccine formulations | Day 0 and Day 28
  Seroconversion is defined as HAI antibody titer < 10 [1/dil] at Day 0 and post-injection titer ≥ 40 [1/dil] at Day 28, or titer ≥ 10 [1/dil] at Day 0 and a ≥ 4-fold increase in titer [1/dil] at Day 28)
2-fold and 4-fold rise in SN antibody titers against each of the H3 antigens | Day 0, Day 7, Day 28, Day 90, Day 180, and Day 365
  Influenza vaccine antibody titers a are measured by SN assay

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (5):
- United States (5):
  - Investigational Site Number 8400003, San Diego, California
  - Investigational Site Number 8400002, Melbourne, Florida
  - Investigational Site Number 8400004, Orlando, Florida
  - Investigational Site Number 8400001, Peoria, Illinois
  - Investigational Site Number 8400005, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: FBP00004 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25266&tenant=MT_SNY_9011